CLINICAL TRIAL: NCT06718140
Title: Personalized Transcranial Focused Ultrasound for Mild Neurocognitive Disorder and Healthy Aging
Brief Title: tFUS for Memory in mNCD and Healthy Adults
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00135826
Record Dates: First submitted 2024-06-11; First posted 2024-12-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Mild Neurocognitive Disorder; Healthy Aging
Keywords: Memory; Mild neurocognitive disorder; Brain stimulation
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: Within-subject crossover between participants; each participant will receive each condition on different days in a counterbalanced order.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Focused Ultrasound to Location A (Experimental): Focused Ultrasound will be administered to location A as condition 1. Stimulation will last 1-10 minutes
  Interventions: Device: Transcranial Focused Ultrasound
- Focused Ultrasound to Location B (Experimental): Focused Ultrasound will be administered to location B as condition 2. Stimulation will last 1-10 minutes
  Interventions: Device: Transcranial Focused Ultrasound
- Focused Ultrasound to Location C (Experimental): Focused Ultrasound will be administered to location C as condition 3. Stimulation will last 1-10 minutes
  Interventions: Device: Transcranial Focused Ultrasound
- Focused Ultrasound to Location D (Sham Comparator): Focused Ultrasound will be administered to location D as condition 4. Stimulation will last 1-10 minutes
  Interventions: Device: Transcranial Focused Ultrasound

INTERVENTIONS:
Device: Transcranial Focused Ultrasound — Using MRI-guided targeting, we will administer focused ultrasound to one of the 4 brain locations

SUMMARY:
Dementia is an ongoing and growing public health crisis in the US and worldwide. The purpose of this study is to examine a form of noninvasive brain stimulation called transcranial focused ultrasound (tFUS) to the hippocampus with the goal of improving memory.

DETAILED DESCRIPTION:
Dementia is an ongoing and growing public health crisis in the US and worldwide. Currently, there are an estimated 6.2 million Americans living with Alzheimer's Disease (AD) the most common form of dementia accounting for roughly 75% of cases. With a growing aging population, this number is estimated to be 13.8 million in the US and 152.8 million people worldwide by 2050 with a 14% lifetime prevalence. It is difficult to treat AD, making it critical to intervene as early as possible. Mild neurocognitive disorder (mNCD) is an early stage of memory and cognitive ability loss that is more severe than normal cognitive decline due to aging. Each year, approximately 15% of people with mNCD develop dementia, making it a critical juncture where intervention could be particularly impactful. Previous research has utilized a novel technique, called transcranial focused ultrasound (tFUS), to change brain function and has measured changes to brain activity through electroencephalography (EEG) using scalp electrodes. This study will apply tFUS to the hippocampus to examine the effects on memory in healthy adults in mNCD.

ELIGIBILITY:
Inclusion Criteria for Healthy Older Adults

* Age 50-85
* English as a first/primary language
* Capacity to consent
* No Diagnosis of mNCD or dementia

Exclusion Criteria for Healthy Older Adults

* Current substance use disorder, bipolar disorder, or schizophrenia spectrum or other psychotic diagnosis
* Daily/weekly anticholinergic or sedative use. Stimulants may be used pending investigator review. Cholinesterase inhibitors, NMDA receptor antagonists, and antidepressants are allowed if on a stable regimen for 4 weeks prior to enrollment
* History of significant or unstable conditions that may impact cognition, such as significant cardiac, cerebrovascular, or metabolic disease, developmental disorder, or other neurologic disease (e.g., moderate to severe TBI, seizures)
* MRI or tFUS contraindications (e.g., metal implants, claustrophobia, conditions or treatments that lower seizure threshold, taking medications that have short half-lives)
* Enrolled in a clinical trial or has received an investigational medication or device in the last 30 days

Inclusion Criteria for mNCD

* Age 50-85
* English as a first/primary language
* Diagnosed with mNCD by a healthcare provider within the past 2 years per NIA-AA or DSM-5 criteria
* Has ≥ 2 impaired scores within one cognitive domain OR ≥ 1 impaired score in ≥ 3 domains, where impaired score is defined as ≤ 16th percentile using demographically-corrected norms
* Must have a co-participant (e.g., spouse, adult child, relative, sibling, cohabitor, friend, or caregiver) with at least weekly in-person contact with the participant

Exclusion Criteria for mNCD

* Prior diagnosis of dementia or major neurocognitive disorder per NIA-AA or DSM-5 criteria, and telephone interview for cognitive status (TICS) score ≤ 22
* Current substance use disorder, bipolar disorder, or schizophrenia spectrum or other psychotic diagnosis
* Daily/weekly anticholinergic or sedative use. Stimulants may be used pending investigator review. Cholinesterase inhibitors, NMDA receptor antagonists, and antidepressants are allowed if on a stable regimen for 4 weeks prior to enrollment
* History of significant or unstable conditions that may impact cognition, such as significant cardiac, cerebrovascular, or metabolic disease, developmental disorder, or other neurologic disease (e.g., moderate to severe TBI, seizures)
* MRI or tFUS contraindications (e.g., metal implants, claustrophobia, conditions or treatments than lower seizure threshold, taking medications that have short half-lives)
* Enrolled in a clinical trial or has received an investigational medication or device in the last 30 days

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Face Name Associative Memory Task (Episodic Memory) effects | Pre- to post-stimulation (within approximately a 1 hour time period)
  Determine the within-subject effects of tFUS on episodic memory (Face Name Associative Memory Task)
Electroencephalography (EEG) effects | Pre- to post-stimulation (within approximately a 1 hour time period)
  Determine the effects of tFUS on EEG recorded from scalp electrodes from pre- to post-stimulation. The investigators will evaluate broadband effects ranging from delta (1-4Hz) to beta (25-40Hz) ranges.

SECONDARY OUTCOMES:
Tolerability of tFUS (self report 0-10 scale) | Pre- to post-stimulation (within approximately a 1 hour time period)
  Ratings on a scale of 0-10 gauging the side effects of stimulation on headache, pain, and other potential side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Caulfield, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States